CLINICAL TRIAL: NCT01247597
Title: DICER1-Related Pleuropulmonary Blastoma Cancer Predisposition Syndrome: A Natural History Study
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110034; 11-C-0034
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12-30

CONDITIONS: Pleuropulmonary Blastoma; Cystic Nephroma; Ovarian Sertoli-Leydig Cell Tumors; Ocular Medulloepithelioma; Nasal Chondromesenchymal Hamartoma
Keywords: Thyroid Cancer; Germline DICER1 Mutation; MicroRNA Biogenesis; Natural History; Pleuropulmonary Blastoma; PPB
MeSH Terms: conditions — Pleuropulmonary blastoma; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: People without pathogenic DICER1 germline variation
- DICER1 (cases): People with pathogenic DICER1 germline variation or history of DICER1-associated tumors

SUMMARY:
Background:

- Pleuropulmonary blastoma (PPB) is a rare fast-growing lung tumor that is associated with other, rare tumor types. Most cases of PPB appear in children younger than 6 years of age. Recently, it has been shown that this condition can be inherited (e.g., mutation of the DICER1 gene). Researchers are studying both clinical and genetic aspects of this newly described condition. They are interested in collecting further medical history and genetic information on individuals and close relatives of individuals who have PPB or other rare associated tumors.

Objectives:

- To study individuals with a personal or a family history of pleuropulmonary blastoma (PPB) or other rare tumors that can be associated with PPB (e.g., cystic nephroma, nasal chondromesenchymal hamartoma, ovarian Sertoli-Leydig cell tumors, ocular medulloepithelioma).

Eligibility:

* Individuals who have been diagnosed with PPB and/or PPB-related tumors.
* Close blood relatives (e.g., parents, siblings, grandparents) of individuals who have been diagnosed with PPB and/or PPB-related tumors.

Design:

* Interested participants can enroll or inquire about this study by calling 1-800-518-8474.
* Participants will be asked to complete family history and medical history questionnaires. They will complete the questionnaire if they are at least 18 years of age, or another person will complete the questionnaire if the key family member is too young to do so on his or her own.
* Participants will be asked to sign a medical record release form to allow researchers to examine detailed medical history information.
* Participants may be asked to have a physical examination and imaging studies, provide blood and saliva samples, or provide tumor tissue from prior biopsies or cancer surgeries.
* Annually, participants will update the family history and individual information questionnaires to document important changes in medical history, and will also update the medical record release form. Participants may be asked to provide additional cheek lining cells and/or blood samples, as well as tumor tissue from any new or planned biopsies or tumor surgeries.
* Treatment will not be provided as part of this protocol.

DETAILED DESCRIPTION:
Study Description:

Multidisciplinary natural history study with self-administered questionnaires, clinical/epidemiologic/genetic evaluations, clinical and research laboratory tests, review of medical records, cancer surveillance, and biospecimen acquisition. In 2009, Hill and colleagues identified heterozygous germline disease-associated variants in DICER1, a gene which encodes a crucial component of the microRNA processing machinery, in patients with familial pleuropulmonary blastoma (PPB). This disorder represents the first reported cancer predisposition syndrome that is due to altered microRNA biogenesis, and its discovery presents a unique and extraordinary opportunity for CGB and DCEG to play a substantial role in the development of this new area, one which is virtually certain to have etiologic ramifications far beyond those related to PPB itself.

Objectives:

1. To establish a cohort of patients with PPB and/or specific neoplasms of the DICER1-related tumor risks (cystic nephroma, nasal chondromesenchymal hamartoma, ovarian Sertoli-Leydig cell and other sex cord-stromal tumors, ocular medulloepithelioma, Wilms tumor, embryonal rhabdomyosarcoma, pineoblastoma, others to be defined), in order to determine the frequency of DICER1 germline disease-associated variants in these patients and their family members. This will also allow us to identify DICER1 disease-associated variant-negative patients who will be crucial for future gene discovery efforts.
2. To characterize the clinical phenotype of, and study the incident and prevalent cancer rates in, these patients and their family members, for all cancers combined, and for each type of cancer, and to identify and confirm the specific types of cancer and benign neoplasms associated with this disorder.
3. To identify differences between patients with a germline disease-associated variant in DICER1 (or another gene(s) from this pathway) who do develop cancer and those who do not develop cancer. These differences may include genotype/phenotype/cancer susceptibility differences, modifier genes (gene-gene interactions) and environmental risk factors (gene-environment interactions). The latter two may be informative for modification of cancer risk in the general population.
4. To develop evidence-based management guidelines for cancer prevention and risk-reduction strategies for patients with PPB and other DICER1-related tumors and their family members prior to and after obtaining answers to the questions/objectives above.
5. To evaluate various parameters related to psychosocial and behavioral issues resulting from being a member of a family at increased risk of PPB and other DICER1-related tumors.
6. To create a biospecimen repository of carefully annotated tissue samples for use in subsequent etiologically-oriented translational research projects. These samples comprise an invaluable resource for current and future studies related to the etiology of, and outcomes following, the various neoplasms that are now known, or later found to be, part of the DICER1-related tumor risk.

Endpoints:

Primary endpoints: include all cancers, with specific attention to those currently thought to be part of the DICER1-related tumor risk.

Secondary endpoints: include non-malignant health issues.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants who meet the eligibility criteria outlined below will be eligible for inclusion in this study regardless of their race, gender, ethnicity, or age.

* Affected individual is defined as:

  * an individual with histologically-confirmed PPB and/or other DICER1-related tumors
  * an individual with a known or suspected DICER1 disease-associated variant
  * an individual from the general population with one or more of the unique tumors of the types associated with DICER1 including (but not exclusively), PPB, cystic nephroma, ovarian Sertoli-Leydig cell and other sex cord-stromal tumors, ocular medulloepithelioma, nasal chondromesenchymal hamartoma, Wilms tumor, embryonal rhabdomyosarcoma, pineoblastoma, pituitary blastoma, ovarian sarcoma, CNS sarcoma and/or thyroid cancer - regardless of their family history. Additional DICER1-related neoplasms may be identified in the future, and they will be added to the protocol as needed.
* Unaffected individual is defined as:

  * a family member (such as parents, siblings, children, or extended family) of an affected participant without a known or suspected DICER1 disease-associated variant or condition and they will be controls.

Other inclusion criteria include:

* All types and amounts of prior therapies are allowed.
* There is no age restriction.
* There is no restriction related to organ and marrow function.
* Ability of the individual or their legal guardian or appropriate surrogate to understand, and their willingness to provide informed consent.

Neonates of affected individuals will be included in the Field Cohort and be eligible for genetic counseling, education, and testing, if indicated and consented by a parent/legal guardian/LAR.

This is entirely a function of meeting the inclusion criteria and not being excluded by the exclusion criteria.

In some instances, patients with histologically-confirmed PPB and/or another neoplasm within the DICER1-related tumor risk and their families will be referred to the Clinical Genetics Branch (CGB) by the International Pleuropulmonary Blastoma (PPB) / DICER1 Registry (IPPBR), provided that the family has previously or currently indicated a desire to be notified of such research opportunities. In non IPPBR cases, the diagnosis will be confirmed by reviewing relevant medical records and relevant surgical pathology material.

EXCLUSION CRITERIA:

Individuals and families referred for evaluation in whom reported diagnoses are not verifiable.

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of patients with PPB and/or specific neoplasms of the PPB spectrum (cystic nephroma, nasal chondromesenchymal hamartoma, ovarian Sertoli-Leydig cell and other sex cord-stromal tumors, ocular medulloepithelioma, Wilms tumor, embryonal rhabdomyosarcoma, pineoblastoma, others to be defined)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-02-13 (Actual)

PRIMARY OUTCOMES:
Psychosocial and Behavioral Issues | On-going
  To evaluate various parameters related to psychosocial and behavioral issues resulting from being a member of a family at increased risk of PPB.
Management Guidelines & Risk-reduction Strategies | On-going
  To develop evidence-based management guidelines for cancer prevention and risk-reduction strategies for PPB patients and their family members prior to and after obtaining answers to the questions/objectives above.
Genetic & Environmental Interactions | On-going
  To identify differences between patients with a germline mutation in DICER1 (or another gene(s) from this pathway) who do develop cancer and those who do not develop cancer. These differences may include genotype/phenotype/cancer susceptibility differences, modifier genes (gene-gene interactions) and environmental risk factors (gene-environment interactions). The latter two may be informative for modification of cancer risk in the general population.
DICER1-Related Pleuropulmonary Blastoma Cancer Predisposition Syndrome | On-going
  To establish a cohort of patients with PPB and/or specific neoplasms of the PPB spectrum (cystic nephroma, nasal chondromesenchymal hamartoma, ovarian Sertoli-Leydig cell and other sex cord-stromal tumors, ocular medulloepithelioma, Wilms tumor, embryonal rhabdomyosarcoma, pineoblastoma, others to be defined), in order to determine the frequency of DICER1 germline mutations in these patients and their family members. This will also allow us to identify DICER1 mutation-negative patients who will be crucial for future gene discovery efforts.
Clinical Phenotype | On-going
  To characterize the clinical phenotype of, and study the incident and prevalent cancer rates in, these patients and their family members, for all cancers combined, and for each type of cancer, and to identify and confirm the specific types of cancer and benign neoplasms associated with this disorder.
Biospecimen Repository | On-going
  To create a biospecimen repository of carefully-annotated tissue samples for use in subsequent etiologically-oriented translational research projects. These samples comprise an invaluable resource for current and future studies related to the etiology of, and outcomes following, the various neoplasms that are now known, or later found to be, part of the PPB syndrome.

SECONDARY OUTCOMES:
Non-tumor phenotypes | On-going
  Secondary endpoints will include characterization of other known or suspected DICER1-related non-tumor health issues such as dysmorphic features, thyroiditis, dental problems, dysmorphology, ophthalmologic abnormalities and pneumothorax. Characterization of individuals and families with DICER1-related non-tumor phenotypes permits identification of people at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Stewart, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - National Cancer Institute - Shady Grove, Rockville, Maryland

REFERENCES:
- [Background] Hill DA, Ivanovich J, Priest JR, Gurnett CA, Dehner LP, Desruisseau D, Jarzembowski JA, Wikenheiser-Brokamp KA, Suarez BK, Whelan AJ, Williams G, Bracamontes D, Messinger Y, Goodfellow PJ. DICER1 mutations in familial pleuropulmonary blastoma. Science. 2009 Aug 21;325(5943):965. doi: 10.1126/science.1174334. Epub 2009 Jun 25. PMID 19556464
- [Background] Manivel JC, Priest JR, Watterson J, Steiner M, Woods WG, Wick MR, Dehner LP. Pleuropulmonary blastoma. The so-called pulmonary blastoma of childhood. Cancer. 1988 Oct 15;62(8):1516-26. doi: 10.1002/1097-0142(19881015)62:83.0.co;2-3. PMID 3048630
- [Background] Hill DA, Jarzembowski JA, Priest JR, Williams G, Schoettler P, Dehner LP. Type I pleuropulmonary blastoma: pathology and biology study of 51 cases from the international pleuropulmonary blastoma registry. Am J Surg Pathol. 2008 Feb;32(2):282-95. doi: 10.1097/PAS.0b013e3181484165. PMID 18223332
- [Derived] Vasta LM, Khan NE, Higgs CP, Harney LA, Carr AG, Harris AK, Schultz KAP, McMaster ML, Stewart DR. Hematologic indices in individuals with pathogenic germline DICER1 variants. Blood Adv. 2021 Jan 12;5(1):216-223. doi: 10.1182/bloodadvances.2020002651. PMID 33570641
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-C-0034.html